CLINICAL TRIAL: NCT00207129
Title: Effect of Capecitabine on the Pharmacokinetics of BMS-247550 on the Pharmacokinetics of Capecitabine and Its Metabolites in Patients With Advanced Malignancies
Brief Title: Effect of Capecitabine on the Pharmacokinetics of BMS-247550 and BMS-247550 on the Pharmacokinetics of Capecitabine and Its Metabolites in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R-Pharm (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA163-038
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Advanced Solid Tumors; Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — ixabepilone; Capecitabine

ARMS (2):
- A (Experimental)
  Interventions: Drug: Ixabepilone
- B (Experimental)
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Ixabepilone — Solution, I.V. infusion, 40 mg/m2, Cycles 1-18: once per cycle (Day 1) cycles 2-18 (6-54 weeks) depending on response.
  Other Names: Ixempra
  Arms: A
Drug: Capecitabine — Tablets, Oral, 1000 mg/m2, Cycle 1: Once (Day 1) Cycle 2: Twice daily (Days 1-5) Cycles 3-18: None, 2 cycles (6 weeks).
  Arms: B

SUMMARY:
The purpose of this study is to test how BMS-247550 (ixabepilone) affects the removal of capecitabine from the body and how capecitabine affects the removal of BMS-247550 from the body.

ELIGIBILITY:
Inclusion Criteria:

* Recovery from surgery or radiation therapy
* Measurable or non-measurable disease
* Available for follow-up

Exclusion Criteria:

* Neuropathy
* Uncontrolled pulmonary or cardiovascular disease
* Known history of HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2004-10; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Effect of capecitabine on the pharmacokinetics of BMS-247550 and to assess the effect of BMS-247550 on the pharmacokinetics of capecitabine

SECONDARY OUTCOMES:
Safety/Tumor response

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, San Antonio, Texas, United States